CLINICAL TRIAL: NCT01179711
Title: The Maximal Tolerable Reduction in Hyperopic Correction in Patients With Refractive Accommodative Esotropia: A 6-month Follow-up Study
Brief Title: Under-correction in Refractive Accommodative Esotropia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Kyung Ah Park, Samsung Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-06-027
Record Dates: First submitted 2010-08-05; First posted 2010-08-11 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Accommodative Esotropia
Keywords: accommodative esotropia
MeSH Terms: interventions — Eyeglasses

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- glasses prescription (Other): At initial visit(of study), the physician will reduce the diopter of hyperopic glasses as much as the patient can maintain their eye alignment (maximum amount 1.5D).
  Interventions: Device: Glasses prescription

INTERVENTIONS:
Device: Glasses prescription — At initial visit(of study), the physician will reduce the diopter of hyperopic glasses as much as the patient can maintain their eye alignment (maximum amount 1.5D).

SUMMARY:
In most clinics, physicians reduce diopter of hyperopic glasses in older patients with accommodative esotropia. However, there are risks of decompensation in that practice. The authors are going to try measure the change of stability of eye alignment after reducing diopter of hyperopic glasses.

DETAILED DESCRIPTION:
Inclusion criteria :

patients with accommodative esotropia

At initial visit(of study), the physician will reduce the diopter of hyperopic glasses as much as the patient can maintain their eye alignment (maximum amount 1.5D).

Outcome measure :

Follow-up examinations are scheduled at 1 week, 1 month, 3 months, and 6 months after the patients begin wearing under-corrected spectacles. At every visit, symptoms such as asthenopia, diplopia, or blurred vision will be documented and ocular examinations, including visual acuity and ocular alignment status for distance and near will be performed. Tests of fusion and stereoacuity will be performed at the 1-month, 3-month, and 6-month follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* patients with accommodative esotropia
* older than 24 months

Exclusion Criteria:

* unstable eye alignment
* older than 18 years

Ages: 24 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
eye alignment | 6 months
  Follow-up examinations are scheduled at 1 week, 1 month, 3 months, and 6 months after the patients begin wearing under-corrected spectacles. At every visit, symptoms such as asthenopia, diplopia, or blurred vision will be documented and ocular examinations including ocular alignment status for distance and near will be performed.

SECONDARY OUTCOMES:
stereopsis | 6 months
  Follow-up examinations are scheduled at 1 week, 1 month, 3 months, and 6 months after the patients begin wearing under-corrected spectacles. At every visit, tests of fusion and stereoacuity will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Sei Yeul Oh, MD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Park KA, Kim SM, Oh SY. The maximal tolerable reduction in hyperopic correction in patients with refractive accommodative esotropia: a 6-month follow-up study. Am J Ophthalmol. 2011 Mar;151(3):535-41.e2. doi: 10.1016/j.ajo.2010.09.023. Epub 2011 Jan 13. PMID 21236414